CLINICAL TRIAL: NCT01871779
Title: The Effect of Different Forms of Exercise on Both the Clinical, Systemic and Local Biological Responses in Intermittent Claudication
Brief Title: Effect of Exercise Training on Protein Expression in Skeletal Muscle Tissue After Exercise in Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flinders University (Other)
Collaborators: Flinders Medical Centre (Other Government); Royal Adelaide Hospital (Other); The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Christopher L Delaney, Doctor, Flinders University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALPAINCLAUD2011
Record Dates: First submitted 2013-05-31; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Treadmill Exercise (Experimental): The first group would undergo standard treadmill exercise to the point of pain and repeat these cycles for a total period of 35-45 minutes twice weekly for 12 weeks
  Interventions: Other: Standard Treadmill Exercise
- Intermittent Treadmill & Resistance Training (Experimental): The second group would have a combination of intermittent treadmill and some resistance training with weights. They will undergo repeated cycles to a maximum of 35-45 minutes twice weekly for 12 weeks
  Interventions: Other: Intermittent treadmill & resistance training

INTERVENTIONS:
Other: Standard Treadmill Exercise — Standard treadmill exercise to the point of pain twice weekly for 35-45 minutes for 12 weeks
  Arms: Standard Treadmill Exercise
Other: Intermittent treadmill & resistance training — Combination of standard treadmill training and resistance training with weights twice weekly for 12 weeks
  Arms: Intermittent Treadmill & Resistance Training

SUMMARY:
Cardiovascular disease remain one of the leading causes of death in Australia, accounting for 47637 (36%) of deaths in 2004.

Peripheral arterial disease (PAD) is a category of cardiovascular disease, characterised by intermittent claudication. This is defined as walking induced pain, cramping, aching, tiredness or heaviness in one or both legs that does not go away with continued walking and is relieved with rest. It is estimated that between 5-10% of individuals aged over 50 years suffer from claudication. The primary and most effective treatment for these patients is focused on improving walking ability and functional status.

Current research has shown that approximately 30% of patients improve with exercise, while 30% continue to deteriorate and the rest show no change. The changes produced at a biochemical and cellular level due to exercise are unknown. To help better understand this, our study will assess the entire range of proteins expressed before and after exercise in the skeletal muscle tissue of patients with intermittent claudication. This will help to identifying key proteins that have a role in improving patient symptoms and outcome.

DETAILED DESCRIPTION:
Why is this clinical problem important?

Peripheral Arterial Disease (PAD) is a major health problem in Australia, with a prevalence of 15% in males aged over 65 years. The direct health care cost of PAD in Australia was $180m in 1994, of which 78% was associated with hospitalisations. PAD is also a marker for advanced cardiovascular disease (CVD) involving coronary, cerebral, renal and aortic vessels; with a 2-3 fold increased risk of CVD-related mortality. In 2006-2007, 25,813 hospitalizations and 2,163 deaths were a result of PAD (Australian Institute of Health and Welfare 2009). The ageing Australian population and the prevalence of PAD increases (Australian Institute of Health and Welfare 2009), the national annual health expenditure on cardiovascular disease is likely to increase, greatly exceeding the 5.4 billion dollars spent in 2000-01 (Australian Bureau of Statistics 2006). The most frequent symptom of mild to moderate PAD is intermittent claudication (IC), defined as walking-induced pain and cramping in one or both legs (most often calves) that is relieved with rest. The primary and most effective treatment for people with intermittent claudication is focused on improving walking ability and functional status.

What is already known about the effect of exercise in intermittent claudication?

The beneficial effects of exercise training as a treatment have been confirmed in several randomised controlled trials. The optimum form of exercise still hasn't been elucidated. The mechanisms of improvement of claudication with exercise are largely unknown. Although exercise stimulates an ischaemic-reperfusion (I-R) insult, repetitive exercise may produce an adaptive response to this I-R insult. Other potential themes include effect of exercise on stimulating or inhibiting angiogenesis and/or muscle protein synthesis.

Although the principal cause of IC is reduced blood flow to the lower limbs relative to increased demand during exercise, the pathophysiology of IC is not completely understood. For example, limb haemodynamics does not closely correlate with clinical presentation or the limitations in peak exercise performance. Haemodynamic measures of the severity of PAD, such as the ankle-brachial systolic blood pressure index (ABI) and blood flow by strain gauge plethysmography, are poor predictors of exercise capacity in patients with IC.

Cross-sectional studies indicate that inflammation is associated with the presence, progression and severity of PAD. This may explain the excess cardiovascular mortality, (at least 50% at 10 years), seen in these patients. The effect of exercise on claudication has been most studied with inflammatory markers in peripheral blood.

What is the importance of measuring protein expression in muscle tissue?

While peripheral blood bio-markers help in understanding the systemic manifestations of claudication, it does not reflect what is happening in the muscles and microcirculation. Most of the changes in protein expression are too subtle to be detected in peripheral blood. The ease of acquisition does not correspond to ease of interrogation. The dynamic range of proteins in serum makes analysis very challenging because high abundance proteins tend to mask those of lower abundance; whilst a small number of proteins including albumin, Beta 2-macroglobulin, transferrin, and immunoglobulins may represent over 90% of serum proteins11.

The protein complement of a cell or tissue is dynamic and reflects the age, life-cycle, and conditions the cell is subjected to or a specific disease state. It is clear that in most diseases, proteins are subjected to numerous changes including post-translational modifications and/or proteolytic cleavage; equally in certain diseases, there is alteration of protein expression. Messenger ribonucleic acid (mRNA) is the molecule encoding the chemical blueprint for a protein. Yet the micro arrays examining differential expression of mRNA will not provide information on post-translational modification, therefore the only way to assess the impact of the proteins is at the protein level.

Some studies have investigated the difference in histochemical and biochemical characteristics of skeletal muscle between patients with PAD and healthy age-matched subjects. Most of the studies into muscle biopsy from patients with PAD have demonstrated alterations in muscle fibre type distribution, denervation and alterations in muscle metabolism with no insight into protein expression12, 13, 14. There is considerable evidence that the metabolic status of skeletal muscle is perturbed in patients with PAD as compared with age-matched healthy controls. Amongst the earliest observations was the unexpected finding that the expression and activity of several mitochondrial enzymes are increased in skeletal muscle from limbs with PAD. The skeletal muscles in patients with IC, do change with exercise but the current evidence does not shed light on the mechanisms of change or if the change is the same in all patients. We do already know that some patients improve with exercise while others do not. A question thus arises as to whether there exists a bio-diversity in these patients' response to exercise.

Armstrong et al studied disturbances in calcium homeostasis of skeletal muscle and suggested that they might play a key role in the development of exercise-induced muscle damage. Some of the immediate muscle changes after exercise have been attributed to protein degradation is initiated by non-lysosomal cysteine proteases, such as calpain. The elevation in intracellular calcium post-exercise can activate the calpains. Muscle tissue expresses three distinct calpains, including the well-characterized ubiquitous calpains - m- calpain, μ-calpain and n-calpain. Wang et al have concluded, in animal studies, that the increased levels of the protease m-calpain, promotes muscle injury whereas the calpastatin protein expression might execute a protective function for muscle injury. This has not yet been investigated in human studies. It can be hypothesised that the levels of calpastatin and m-calpain are important in explaining the variable response to exercise in IC and why some patients improve and others do not.

There is some conflicting evidence on the benefit of exercise. Tsai et al have found that the normal training effect on the glucose transporter 4 (GLUT4) gene expression was completely eliminated by both acute and chronic ischemia at the pre-translational level. In addition, the chronic ischemia-induced muscle atrophy was seen to be more severe in the exercise-trained rats than in the untrained rats. This result suggests that for individuals with impaired microvascular conditions, exercise training might not be beneficial in maintaining muscle mass. Thus the effect of exercise training in human subjects with IC (ischaemia) is yet to be elucidated.

We know that all subjects differ in their capacity for exercise and patients with intermittent claudication are no different. Patients undergoing exercise for intermittent claudication, would be different in terms of their expression of proteins due to exercise. For this reason, patients would act as their own controls by means of a biopsy from an unaffected muscle of each individual.

An open ended mass spectroscopy examination of proteins in the exercising skeletal muscle would give an insight into the mechanistic pathway of the exercise effect in intermittent claudication.

What is the relation between protein expression and inflammation in the exercise with intermittent claudication?

The clinical model of exercise inducing an ischaemia-reperfusion type injury has been substantiated by evidence of markers of inflammation. Neutrophils are the first cells to begin accumulating in the tissue at the injury site, destroying necrotic tissue through phagocytosis while working in conjunction with resident macrophages from the muscle tissue itself. Neutrophil presence has been documented in muscle after various types of eccentric exercise. A study looking at neutrophil function in exercising claudicants showed increased neutrophil activation manifest by increased expression of the neutrophil adhesion receptor cluster of differentiation antigen IIb (CD11b) and degranulation manifest by an increase in plasma neutrophil elastase. This occurred immediately after exercise in these patients with intermittent claudication. Whether this equates to a trend to predict outcomes is still not clear.

The protease m-Calpain is chemotactic factor for neutrophils and may play a role in the local and systemic inflammatory response. Such adaptations in cellular inflammatory responses have been reported earlier by Kunimatsu et al. Together with Calpastatin, these proteins may hold a key in the link between local muscle damage, repair and inducing a systemic inflammatory response.

Chemical modification of proteins may play a role in the pathogenesis of disorders ranging from diabetes to atherosclerosis and ischemia-reperfusion injury and perhaps to the aging process itself. Advanced Glycosylation End products (AGEs) are the end products of glycosylation reactions in which a sugar molecule bonds to either a protein or lipid molecule without an enzyme to control the reaction. The formation and accumulation of AGEs has been implicated in the progression of age related disease, in particular cardiovascular disease. They have a range of pathological effects, including inhibition of vascular dilatation by interfering with nitric oxide (Endothelium Derived Relaxation factor), binding macrophage and endothelial cells to induce the secretion of inflammatory cytokines and enhancing oxidative stress. We hypothesise that exercise stimulates glucose uptake by the endothelial cells increasing the synthesis of AGE's. It remains to be determined whether exercise again enhances or reduces this process.

The aim of this study is to examine inflammatory biomarkers, including Interleukin-6 (IL-6), Neutrophil elastase and Advanced Glycated End-products with proteins known to influence tissue damage or repair (Calpains and Calpastatin) to determine the effect of different forms of exercise on this process, in order to determine

1. Is exercise appropriate for all patients? i.e.

   1. Do all patients respond with a pro inflammatory response? and
   2. Does exercise produce an adaptive response to this in all patients? or
   3. Does exercise stimulate an I-R insult in some patients that is not reduced by exercise training?
   4. What is the local tissue response to exercise in terms of tissue damage or repair (as measured by protein analysis)
2. What is the best form of exercise for these suitable patients?
3. Is there a biodiversity in patients' response to exercise in terms of

   1. Systemic inflammatory response (based on IL-6, Neutrophil Elastase & AGE's)?
   2. Local response (based on protein analysis)?
4. Does the physiological response to exercise in these patients reduce the risk of CVD related morbidity/mortality?

   a. As evidenced by changes in cardiopulmonary exercise testing (CPET) outcome parameters and endothelial function.
5. Is impaired endothelial function reversible? a. As measured by flow-mediated dilatation.

The combined use of data from systemic blood and local muscle tissue would help to characterise the metabolic and functional consequences of age associated PAD changes in skeletal muscle. It would also help to identify a mechanistic pathway by which exercise exerts its effect on the patient with intermittent claudication.

ELIGIBILITY:
Inclusion Criteria:

1. All claudicants with a walking distance of 50 metres or more with a resting ankle brachial index equal to or less than 0.9.
2. Claudicants meeting above criteria, who may have previously had a percutaneous arterial intervention for symptom control more than 12 months ago.

Exclusion Criteria:

1. Patients with lower limb pain of other aetiologies - neurogenic claudication evidenced by normal ankle brachial indices and duplex ultrasound.
2. Patients with lower limb ischaemic rest pain
3. Patients with current or previous tissue loss, such as ulcers or necrotic lesions.
4. Patients with recent (<12 months) history of peripheral vascular interventions for symptoms.
5. Patients with pre-existing cardiac or respiratory problems limiting exercise.
6. Patients with previous disabling strokes which would restrict exercise regimes
7. Patients with anticoagulation or blood dyscrasias.
8. Women who are pre-menopausal,
9. Women receiving hormone-replacement therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Improvement in Pain Free Walking Distance | Change from baseline (pre intervention) to 12 weeks (post intervention)
  Patients will be exercised based on standard protocols and monitored for improvements in Maximal walking distance and Pain Free Walking distances.

SECONDARY OUTCOMES:
Skeletal muscle protein expression | Change from baseline (pre intervention) to 12 weeks (post intervention)
  Skeletal muscle samples obtained from ultrasound guided biopsy of symptomatic medial gastrocnemius muscle will be assessed for protein activity of proteins from the calpain family, specifically, m-calpain and calpastatin.
Inflammatory cytokines | Change from baseline (pre intervention) to 12 weeks (post intervention)
  Fasting C Reactive Protein, Interleukin 6 and Neutrophil Elastase will be analysed from serum via enzyme-linked immunosorbent assays.
Endothelial function | Change from baseline (pre intervention) to 12 weeks (post intervention)
  Endothelium-mediated changes in vascular tone will be quantified by reactive hyperemia-peripheral artery tonometry index and flow-mediated dilatation using high resolution ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Delaney, BMBS, Principal Investigator — Flinders University and Flinders Medical Centre Department of Vascular Surgery; James I Spark, MBChB, MD,, Principal Investigator — Flinders University and Flinders Medical Centre Department of Vascular Surgery
Locations (1):
- Repatriation General Hospital, Daw Park, South Australia, Australia

REFERENCES:
- [Derived] Delaney CL, Miller MD, Dickinson KM, Spark JI. Change in dietary intake of adults with intermittent claudication undergoing a supervised exercise program and compared to matched controls. Nutr J. 2014 Oct 15;13:100. doi: 10.1186/1475-2891-13-100. PMID 25316347